CLINICAL TRIAL: NCT06860854
Title: The Effect of Epidural Analgesia on Uterine Contractility and Intrapartum Fetal Well-being - Study Protocol for a Prospective Observational Study "EPI-CARE"
Brief Title: EPidural's Impact on Contractions and Fetal REsponse
Acronym: EPI-CARE
Status: Not yet recruiting | Type: Observational
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Król Joanna, Principal Investigator, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Other Study IDs: EPI-CARE ver. 1
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Epidural Anesthesia in Labor and Delivery; Doppler Ultrasound; Uterine Contraction
Keywords: Epidural Analgesia; Uterine Contractility; Maternal-Fetal Hemodynamics; Cardiotocography (CTG) Patterns
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients in Labor: The study aims to recruit 200 patients in spontaneous or induced labor at 37-42 weeks of gestation, requesting the epidural labor analgesia (ELA) and meeting the inclusion criteria.
  Interventions: Procedure: Epidural Analgesia

INTERVENTIONS:
Procedure: Epidural Analgesia — The eligible patients will have their vital signs (blood pressure, saturation, heart rate) and the Doppler velocities in the uterine arteries, umbilical artery and the fetal middle cerebral artery measured directly before the administration of ELA. They will be also asked to rate their level of pain on the visual analogue scale (VAS).
  The specific method and drug regimen for ELA will be determined by the attending anesthesiologist. The mode of administration (continuous infusion, intermittent bolus, or patient-controlled epidural analgesia) will be recorded along with the anesthetic agents used for future subgroup analysis.
  The vital signs, the Doppler velocities and VAS score will be recorded after 30, 60 and 120 minutes. After 2 hours the patients will be examined to assess the progress of labor.

SUMMARY:
This prospective observational study aims to assess the impact of epidural analgesia (ELA) on uterine contractility, cardiotocography (CTG) patterns, and maternal-fetal hemodynamics in term pregnancies. The study will recruit 200 laboring patient receiving ELA and evaluate changes in uterine contractions, Doppler blood flow parameters, and fetal heart rate tracings before and after ELA administration. Secondary analyses will compare outcomes between primiparous and multiparous women, as well as between uncomplicated and complicated pregnancies. Pain relief effectiveness will be correlated with observed changes. This study will provide a comprehensive understanding of ELA's effects on labor progression and fetal well-being, addressing gaps in existing research.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* singleton pregnancy
* signed informed consent form
* patients in labor
* cervical dilation ≥ 3cm,
* patient requesting and eligible for epidural analgesia
* normal CTG trace for at least 30 minutes before epidural analgesia

Exclusion Criteria:

* < than 18 years old
* preterm delivery
* labor induced or stimulated by oxytocin
* multiple pregnancy
* fetal malformations
* < than 3cm cervical dilation
* lack of CTG trace for at least 30 minutes before epidural analgesia
* patient not requesting or not eligible for epidural analgesia
* informed consent form not signed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient in labor admitted to the Clinical Department of Obstetrics and Perinatology at the National Medical Institute of the Ministry of the Interior and Administration in Warsaw, Poland and meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in uterine contractility | From enrollment to 120 minutes after the administration of epidural analgesia
  Uterine activity will be monitored using the external tocography and expressed as number of contractions per 10 minutes.
  Due to known limitations of the external tocography the labor progression, defined as the change in cervical dilation between the two vaginal examinations (the patients will be examined just before the administration of epidural analgesia and two hours after) will also be recorded in cm.
Changes in maternal and fetal doppler velocities | From enrollment to 24 hours after labor
  The pulsatility index (PI) of maternal uterine arteries, umbilical artery and fetal middle cerebral artery will be assessed by ultrasound before and 30, 60 and 120 minutes after the administration of epidural analgesia. Additionally, the PI in maternal uterine artery will be measured within first 24 hours after labor.
Changes in cardiotocography (CTG) patterns | From enrollment up to 120 minutes after the administration of epidural
  CTG patterns will be monitored using the external tocography. The change in CTG patterns after the administration of epidural analgesia will be assessed by experts overlooking the study and they will be labeled as normal, suspicious or pathological using the FIGO guidelines.

SECONDARY OUTCOMES:
Differences between primiparous and multiparous patients | From enrollment to 120 minutes after the administration of ELA
  The primary outcomes will be compared between primiparous and multiparous patients with the use of subgroup analyses.
Differences between complicated and uncomplicated pregnancies | From enrollment up to 120 minutes after the administration of ELA
  The subgroup analyses will help to determine whether the changes in primary outcomes differ between normal pregnancies and those complicated with diabetes mellitus, hypertension etc.
The correlation of pain relief with changes in uterine contractility and maternal-fetal hemodynamics | From the enrollment up to 120 minutes after the administration of ELA
  The pain relief will be measured comparing the difference between scores on the visual analog scale (VAS) from 0 (no pain) to 10 (worst pain possible) before and after the use of epidural analgesia. Then using the primary outcomes we will study whether the pain relief correlates with the changes in uterine contractility and maternal-fetal doppler velocities.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Department of Obstetrics and Perinatology at the National Medical Institute of the Ministry of the Interior and Administration, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided